CLINICAL TRIAL: NCT02538666
Title: A Randomized, Multicenter, Double-Blind, Phase 3 Study of Nivolumab, Nivolumab in Combination With Ipilimumab, or Placebo as Maintenance Therapy in Subjects With Extensive-Stage Disease Small Cell Lung Cancer (ED-SCLC) After Completion of Platinum-based First Line Chemotherapy (CheckMate 451: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 451)
Brief Title: An Investigational Immuno-therapy Study of Nivolumab, or Nivolumab in Combination With Ipilimumab, or Placebo in Patients With Extensive-Stage Disease Small Cell Lung Cancer (ED-SCLC) After Completion of Platinum-based Chemotherapy
Acronym: CheckMate 451
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-451; 2015-002441-61 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab monotherapy (Experimental): Nivolumab intravenous fusion
  Interventions: Biological: Nivolumab
- Nivolumab and ipilimumab combination therapy (Experimental): Nivolumab and ipilimumab intravenous fusion
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Nivolumab
  Other Names: Opdivo
  Arms: Nivolumab and ipilimumab combination therapy; Nivolumab monotherapy
Biological: Ipilimumab
  Other Names: Yervoy
  Arms: Nivolumab and ipilimumab combination therapy
Other: Placebo
  Arms: Placebo

SUMMARY:
In this study, all patients must have already completed first-line chemotherapy to treat extensive-stage disease small cell lung cancer. The purpose of this study is to show that nivolumab, or nivolumab plus ipilimumab followed by nivolumab by itself, will prolong overall survival when administered as consolidation treatment in patients that are stable or responding after chemotherapy. Patients receiving treatment will be compared with patients taking placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed extensive stage disease SCLC
* Ongoing response of stable disease or better following 4 cycles of platinum-based first line chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Subjects with symptomatic Central Nervous System (CNS) metastases
* Subjects receiving consolidative chest radiation
* Subjects with active, known, or suspected autoimmune disease are excluded
* All side effects attributed to prior anti-cancer therapy must have resolved to Grade 1 or baseline

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (195):
- United States (28):
  - Local Institution - 0003, Sacramento, California
  - Local Institution - 0202, New Haven, Connecticut
  - Local Institution - 0127, Fort Myers, Florida
  - Local Institution - 0007, Jacksonville, Florida
  - Local Institution - 0128, St. Petersburg, Florida
  - Local Institution - 0010, Atlanta, Georgia
  - Local Institution - 0013, Indianapolis, Indiana
  - Local Institution - 0061, Fairway, Kansas
  - Local Institution - 0012, Wichita, Kansas
  - Local Institution - 0032, Lexington, Kentucky
  - Local Institution - 0051, Baltimore, Maryland
  - Local Institution - 0107, Boston, Massachusetts
  - Local Institution - 0207, Boston, Massachusetts
  - Local Institution - 0015, St Louis, Missouri
  - Local Institution - 0008, New York, New York
  - Local Institution - 0014, Durham, North Carolina
  - Local Institution - 0016, Winston-Salem, North Carolina
  - Local Institution - 0215, Fargo, North Dakota
  - Local Institution - 0129, Cincinnati, Ohio
  - Local Institution - 0009, Columbus, Ohio
  - Local Institution - 0001, Portland, Oregon
  - Local Institution - 0034, Portland, Oregon
  - Local Institution - 0004, Allentown, Pennsylvania
  - Local Institution - 0002, Sayre, Pennsylvania
  - Local Institution - 0005, Charleston, South Carolina
  - Local Institution - 0213, Sioux Falls, South Dakota
  - Local Institution - 0011, Salt Lake City, Utah
  - Local Institution - 0006, Richmond, Virginia
- Argentina (5):
  - Local Institution - 0110, Berazategui, Buenos Aires
  - Local Institution - 0088, Capital Federal, Buenos Aires
  - Local Institution - 0109, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution - 0188, Córdoba
  - Local Institution - 0029, San Miguel de Tucumán
- Australia (6):
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Wollongong, New South Wales
  - Local Institution, Birtinya, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Local Institution - 0137, Adelaide, South Australia
  - Local Institution - 0035, East Melbourne, Victoria
- Austria (3):
  - Local Institution - 0174, Innsbruck
  - Local Institution - 0173, Salzburg
  - Local Institution - 0172, Vienna
- Belgium (3):
  - Local Institution - 0057, Brussels
  - Local Institution - 0059, Charleroi
  - Local Institution - 0060, Roeselare
- Brazil (8):
  - Local Institution - 0067, Fortaleza, Ceará
  - Local Institution - 0068, Belo Horizonte, Minas Gerais
  - Local Institution - 0063, Ijuí, Rio Grande do Sul
  - Local Institution - 0064, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0017, Itajaí, Santa Catarina
  - Local Institution - 0081, Barretos, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, Salvador
- Canada (5):
  - Local Institution - 0094, Edmonton, Alberta
  - Local Institution - 0136, Moncton, New Brunswick
  - Local Institution - 0102, Greater Sudbury, Ontario
  - Local Institution - 0123, Oshawa, Ontario
  - Local Institution - 0111, Windsor, Ontario
- China (19):
  - Local Institution - 0238, Hefei, Anhui
  - Local Institution - 0243, Hefei, Anhui
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution - 0221, Harbin, Heilongjiang
  - Local Institution - 0244, Wuhang, Hubei
  - Local Institution - 0248, Nantong, Jiangsu
  - Local Institution - 0230, Nanchang, Jiangxi
  - Local Institution, Changchun, Jilin
  - Local Institution - 0237, Shenyang, Liaoning
  - Local Institution - 0220, Shanghai, Shanghai Municipality
  - Local Institution - 0228, Shanghai, Shanghai Municipality
  - Local Institution - 0233, Shanghai, Shanghai Municipality
  - Local Institution - 0245, Shanghai, Shanghai Municipality
  - Local Institution - 0232, Kunming, Yunnan
  - Local Institution - 0239, Hangzhou, Zhejiang
  - Local Institution - 0227, Hangzhou, Zhejiang
  - Local Institution - 0246, Wenzhou, Zhejiang
  - Local Institution - 0247, Changsha
  - Local Institution - 0240, Guangzhou
- Colombia (3):
  - Local Institution, Montería, Departamento de Córdoba
  - Local Institution - 0078, Bogotá
  - Local Institution, Medellín
- Finland (4):
  - Local Institution - 0044, Oulu
  - Local Institution - 0043, Tampere
  - Local Institution - 0045, Turku
  - Local Institution - 0046, Vaasa
- France (9):
  - Local Institution - 0149, Strasbourg, Alsace
  - Local Institution - 0208, Avignon Cedes 9
  - Local Institution - 0099, Lyon
  - Local Institution - 0098, Marseille
  - Local Institution - 0097, Paris
  - Local Institution - 0095, Pierre-Bénite
  - Local Institution - 0100, Rennes
  - Local Institution - 0150, Saint-Herblain
  - Local Institution - 0096, Toulouse
- Germany (8):
  - Local Institution - 0171, Augsburg
  - Local Institution - 0170, Bad Berka
  - Local Institution - 0168, Berlin
  - Local Institution - 0164, Bochum
  - Local Institution - 0166, Gauting
  - Local Institution - 0165, Großhansdorf
  - Local Institution - 0169, Immenhausen
  - Local Institution - 0167, Tübingen
- Greece (2):
  - Local Institution - 0080, N.Kifissia
  - Interbalkan European Medical Center, Thessaloniki
- Local Institution - 0052, Hong Kong, Hong Kong
- Ireland (5):
  - Local Institution - 0161, Wilton, CORK
  - Local Institution - 0175, Dublin
  - Local Institution, Dublin
  - Local Institution - 0162, Galway
  - Local Institution - 0214, Limerick
- Israel (5):
  - Local Institution, Haifa
  - Local Institution - 0093, Jerusalem
  - Local Institution, Petah Tikva
  - Local Institution - 0090, Tel Aviv
  - Local Institution - 0089, Ẕerifin
- Italy (5):
  - Local Institution - 0027, Milan, Lombardy
  - Local Institution - 0026, Avellino
  - Local Institution - 0025, Bologna
  - Local Institution - 0112, Messina
  - Local Institution - 0082, Perugia
- Japan (22):
  - Local Institution - 0139, Kashiwa-shi, Chiba
  - Local Institution - 0142, Matsuyama, Ehime
  - Local Institution - 0146, Fukuoka, Fukuoka
  - Local Institution - 0200, Kurume-shi, Fukuoka
  - Local Institution - 0198, Gifu, Gifu
  - Local Institution - 0143, Sapporo, Hokkaido
  - Local Institution - 0076, Kobe, Hyōgo
  - Local Institution - 0138, Kanazawa, Ishikawa-ken
  - Local Institution - 0072, Yokohama, Kanagawa
  - Local Institution - 0070, Sendai, Miyagi
  - Local Institution - 0069, Sendai, Miyagi
  - Local Institution - 0077, Kurashiki-shi, Okayama-ken
  - Local Institution, Hirakata-shi, Osaka
  - Local Institution - 0145, Osaka, Osaka
  - Local Institution - 0075, Osaka-sayama-shi, Osaka
  - Local Institution - 0083, Takatsuki-shi, Osaka
  - Local Institution - 0193, Hidaka, Saitama
  - Local Institution - 0141, Bunkyo-ku, Tokyo
  - Local Institution - 0071, Chuo-ku, Tokyo
  - Local Institution - 0140, Koto-ku, Tokyo
  - Local Institution - 0144, Shinjuku-ku, Tokyo
  - Local Institution - 0216, Wakayama
- Mexico (4):
  - Local Institution - 0020, León, Guanajuato
  - Local Institution - 0019, Mexico City, Mexico City
  - Local Institution - 0028, Monterrey, Nuevo León
  - Local Institution - 0135, Querétaro
- Netherlands (3):
  - Local Institution - 0158, 's-Hertogenbosch
  - Local Institution, Eindhoven
  - Local Institution - 0159, Rotterdam
- Peru (2):
  - Local Institution, Miraflores, Lima region
  - Local Institution, Lima
- Poland (4):
  - Local Institution - 0041, Gdansk
  - Local Institution - 0054, Gdynia
  - Local Institution - 0053, Olsztyn
  - Local Institution - 0187, Warsaw
- Romania (6):
  - Local Institution - 0199, Bucharest
  - Local Institution - 0186, Bucharest
  - Local Institution - 0182, Craiova
  - Local Institution - 0178, Lasi
  - Local Institution - 0212, Romania
  - Local Institution - 0181, Timisoara, Timis
- Russia (6):
  - Local Institution - 0148, Moscow
  - Local Institution - 0217, Moscow
  - Local Institution - 0209, Moscow
  - Local Institution - 0116, Saint Petersburg
  - Local Institution - 0157, Saint Petersburg
  - Local Institution - 0115, Saint Petersburg
- Local Institution - 0050, Singapore, Singapore
- South Africa (4):
  - Local Institution - 0087, Sandton, Gauteng
  - Local Institution - 0084, Cape Town, Western Cape
  - Local Institution - 0085, Cape Town, Western Cape
  - Local Institution - 0086, George, Western Cape
- South Korea (5):
  - Local Institution - 0047, Seongnam-si, Gyeonggi-do
  - Local Institution - 0024, Suwon, Kyǒnggi-do
  - Local Institution - 0021, Gangnam-gu
  - Local Institution - 0022, Seoul
  - Local Institution - 0154, Seoul
- Spain (5):
  - Local Institution - 0132, Barcelona
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Seville
- Sweden (2):
  - Local Institution - 0124, Lund
  - Local Institution - 0185, Uppsala
- Switzerland (3):
  - Local Institution - 0179, Aarau
  - Local Institution - 0180, Geneva
  - Local Institution - 0191, Sankt Gallen
- Taiwan (2):
  - Local Institution - 0049, Tainan, TNN
  - Local Institution - 0048, Taoyuan District
- United Kingdom (7):
  - Local Institution - 0153, Truro, Cornwall
  - Local Institution - 0118, London, Greater London
  - Local Institution - 0201, London, Greater London
  - Local Institution - 0121, Metropolitan Borough of Wirral, Lancashire
  - Local Institution - 0152, Oxford, Oxfordshire
  - Local Institution - 0151, Sutton, Surrey
  - Local Institution - 0192, Sheffield

REFERENCES:
- [Derived] Kang YK, Reck M, Nghiem P, Feng Y, Plautz G, Kim HR, Owonikoko TK, Boku N, Chen LT, Lei M, Chang H, Lin WH, Roy A, Bello A, Sheng J. Assessment of hyperprogression versus the natural course of disease development with nivolumab with or without ipilimumab versus placebo in phase III, randomized, controlled trials. J Immunother Cancer. 2022 Apr;10(4):e004273. doi: 10.1136/jitc-2021-004273. PMID 35383114
- [Derived] Owonikoko TK, Park K, Govindan R, Ready N, Reck M, Peters S, Dakhil SR, Navarro A, Rodriguez-Cid J, Schenker M, Lee JS, Gutierrez V, Percent I, Morgensztern D, Barrios CH, Greillier L, Baka S, Patel M, Lin WH, Selvaggi G, Baudelet C, Baden J, Pandya D, Doshi P, Kim HR. Nivolumab and Ipilimumab as Maintenance Therapy in Extensive-Disease Small-Cell Lung Cancer: CheckMate 451. J Clin Oncol. 2021 Apr 20;39(12):1349-1359. doi: 10.1200/JCO.20.02212. Epub 2021 Mar 8. PMID 33683919
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 907 participants were randomized and 903 were treated. 2 participants were in both the Global and China population.
Groups:
- Placebo: 100 mL of 0.9% Sodium Chloride Solution or 5% Dextrose administered as placebo for nivolumab and ipilimumab as an IV infusion
- Nivolumab 240 mg: Nivolumab 240 mg administered every 2 weeks as a 30-minute IV infusion
- Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg: Nivolumab 1 mg/kg (30-minute IV infusion) + Ipilimumab 3 mg/kg (90-minute IV infusion) administered every 3 weeks for 4 doses, followed by nivolumab 240 mg every 2 weeks
Period: Pre-Treatment
Arm/Group | Placebo | Nivolumab 240 mg | Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Started (Started = Randomized) | 300 | 304 | 303
Global | 275 | 280 | 279
China | 26 | 25 | 24
Completed (Completed = Treated) | 298 | 303 | 302
Not Completed | 2 | 1 | 1
Not completed — Disease progression | 1 | 0 | 0
Not completed — no longer meets study criteria | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 1
Period: Treatment
Arm/Group | Placebo | Nivolumab 240 mg | Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Started (Started = Started Treatment) | 298 | 303 | 302
Global | 273 | 279 | 278
China | 26 | 25 | 24
Completed (Completed = Continuing in treatment period) | 0 | 0 | 0
Not Completed | 298 | 303 | 302
Not completed — Disease progression | 270 | 227 | 165
Not completed — Study drug toxicity | 1 | 29 | 92
Not completed — Death | 0 | 2 | 3
Not completed — Adverse event unrelated to study drug | 8 | 10 | 15
Not completed — Participant request to discontinue study treatment | 3 | 6 | 11
Not completed — Participant withdrew consent | 2 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Maximum clinical benefit | 4 | 3 | 4
Not completed — Poor/non-compliance | 0 | 1 | 0
Not completed — Participant no longer meets study criteria | 0 | 2 | 0
Not completed — Administrative reason by sponsor | 0 | 0 | 1
Not completed — Other reasons | 8 | 15 | 5
Not completed — Not reported | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nivolumab 240 mg | Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | Total
Number analyzed (Participants) | 300 | 304 | 303 | 907
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 161 | 149 | 152 | 462
  ≥ 65 and < 75 | 113 | 120 | 115 | 348
  ≥ 75 and < 85 | 26 | 35 | 35 | 96
  ≥ 85 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 105 | 101 | 309
  Male | 197 | 199 | 202 | 598
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 15 | 40
  Not Hispanic or Latino | 160 | 164 | 171 | 495
  Unknown or Not Reported | 126 | 129 | 117 | 372
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 94 | 82 | 82 | 258
  Black or African American | 2 | 6 | 1 | 9
  White | 198 | 213 | 216 | 627
  Other | 6 | 3 | 3 | 12
  Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of Nivolumab + Ipilimumab Versus Placebo In The Global Population
Description: OS was defined as the time from randomization to the date of death. A participant who had not died was censored at last known alive date. OS was followed up during the blinded study drug treatment and every 3 months via in-person or phone contact after participant discontinued the blinded study drug
Time Frame: From randomization to 400 deaths across the two treatment groups (Nivo+Ipi vs Placebo) (up to approximately 37 months)
Population: All randomized participants in the nivolumab + ipilimumab and placebo arms in the global population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Global Placebo: 100 mL of 0.9% Sodium Chloride Solution or 5% Dextrose administered as placebo for nivolumab and ipilimumab as an IV infusion
- Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg: Nivolumab 1 mg/kg (30-minute IV infusion) + Ipilimumab 3 mg/kg (90-minute IV infusion) administered every 3 weeks for 4 doses, followed by nivolumab 240 mg every 2 weeks
Arm/Group | Global Placebo | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 275 | 279
Months | 9.56 [8.18 to 11.01] | 9.17 [8.15 to 10.25]
Statistical Analysis 1: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; nivolumab + ipilimumab over placebo; Test type: Superiority; p = 0.3693, Stratified Log Rank; Stratified by response to ECOG PS (0vs1), gender (MvF), irradiation following chemotherapy (YorN) as entered in IVRS; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.75 to 1.12] — based on stratified 3-arms Cox proportional hazard model

2. Secondary Outcome: Overall Survival (OS) of Nivolumab Versus Placebo
Description: Overall Survival (OS) comparing nivolumab monotherapy versus placebo. OS was defined as the time from randomization to the date of death. A participant who had not died was censored at last known alive date. OS was followed up during the blinded study drug treatment and every 3 months via in-person or phone contact after participant discontinued the blinded study drug.
Time Frame: From randomization to the date of death or last known alive date (up to approximately 73 months)
Population: All randomized participants in the nivolumab monotherapy and placebo arms
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Global Nivolumab 240 mg; China Nivolumab 240 mg: Nivolumab 240 mg administered every 2 weeks as a 30-minute IV infusion
- China Placebo: 100 mL of 0.9% Sodium Chloride Solution or 5% Dextrose administered as an IV infusion
Arm/Group | Global Placebo | Global Nivolumab 240 mg | China Placebo | China Nivolumab 240 mg
Number analyzed (Participants) | 275 | 280 | 26 | 25
Months | 9.56 [8.18 to 11.01] | 10.18 [9.43 to 11.99] | 9.28 [5.59 to 14.26] | 8.18 [7.20 to 14.26]
Statistical Analysis 1: Comparison: Global Placebo vs Global Nivolumab 240 mg; Global nivolumab over global placebo; Test type: Superiority; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.68 to 0.97] — Hazard Ratios are based on stratified 3-arms Cox proportional hazard model
Statistical Analysis 2: Comparison: China Placebo vs China Nivolumab 240 mg; China nivolumab over China Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.53 to 1.66] — Hazard Ratios are based on unstratified 3-arms Cox proportional hazard model

3. Secondary Outcome: Overall Survival (OS) of Nivolumab + Ipilimumab Versus Nivolumab
Description: Overall Survival (OS) comparing Nivolumab + Ipilimumab Versus Nivolumab. OS was defined as the time from randomization to the date of death. A participant who had not died was censored at last known alive date. OS was followed up during the blinded study drug treatment and every 3 months via in-person or phone contact after participant discontinued the blinded study drug.
Time Frame: From randomization to the date of death or last known alive date (up to approximately 73 months)
Population: All randomized participants in the Nivolumab + Ipilimumab and Nivolumab arms
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg: Nivolumab 1 mg/kg (30-minute IV infusion) + Ipilimumab 3 mg/kg (90-minute IV infusion) administered every 3 weeks for 4 doses, followed by nivolumab 240 mg every 2 weeks
Arm/Group | Global Nivolumab 240 mg | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | China Nivolumab 240 mg | China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 280 | 279 | 25 | 24
Months | 10.18 [9.43 to 11.99] | 9.17 [8.15 to 10.35] | 8.18 [7.20 to 14.26] | 10.48 [7.13 to 13.40]
Statistical Analysis 1: Comparison: Global Nivolumab 240 mg vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg vs China Nivolumab 240 mg; Global nivolumab + ipilimumab over global nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.94 to 1.36] — Hazard Ratios are based on stratified 3-arms Cox proportional hazard model
Statistical Analysis 2: Comparison: China Nivolumab 240 mg vs China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; China nivolumab + ipilimumab over China nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.56 to 1.79] — Hazard Ratios are based on unstratified 3-arms Cox proportional hazard model

4. Secondary Outcome: Progression Free Survival (PFS) Per BICR
Description: PFS was defined as the time between the date of randomization and the first date of documented progression as determined by Blind Independent Central Review (BICR) or death due to any cause, whichever occurred first. Participants who died with no reported progression were considered to have progressed on the date of death. Participants who did not progress or die were censored on the date of their last evaluable tumor assessment on or prior to initiation of the subsequent anti-cancer therapy. Participants who did not have any on study tumor assessments and did not die (or died after initiation of the subsequent anti- cancer therapy) were censored on their date of randomization. Participants who started any subsequent anti- cancer therapy without a prior reported Progressive Disease (PD) per BICR were censored at the last evaluable tumor assessment on or prior to initiation of the subsequent anti-cancer therapy.
Time Frame: From randomization to the date of the first documented tumor progression or death due to any cause (up to approximately 73 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Global Placebo | Global Nivolumab 240 mg | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | China Placebo | China Nivolumab 240 mg | China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 275 | 280 | 279 | 26 | 25 | 24
Months | 1.41 [1.41 to 1.48] | 1.94 [1.61 to 2.63] | 1.74 [1.48 to 2.63] | 1.38 [1.28 to 2.56] | 1.58 [1.38 to 4.11] | 1.54 [1.28 to 2.73]
Statistical Analysis 1: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; Global nivolumab + ipilimumab over global placebo; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.62 to 0.88] — Hazard Ratios are based on stratified 3-arms Cox proportional hazard model
Statistical Analysis 2: Comparison: Global Placebo vs Global Nivolumab 240 mg; Global nivolumab over global placebo; Test type: Superiority; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.55 to 0.79] — Hazard Ratios are based on stratified 3-arms Cox proportional hazard model
Statistical Analysis 3: Comparison: Global Nivolumab 240 mg vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; Global nivolumab+ ipilimumab over nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.94 to 1.35] — Hazard Ratios are based on stratified 3-arms Cox proportional hazard model
Statistical Analysis 4: Comparison: China Placebo vs China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; China Nivolumab + Ipilimumab over China placebo; Test type: Superiority; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.33 to 1.12] — Hazard Ratios are based on unstratified 3-arms Cox proportional hazard model
Statistical Analysis 5: Comparison: China Placebo vs China Nivolumab 240 mg; China Nivolumab over China placebo; Test type: Superiority; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.24 to 0.85] — Hazard Ratios are based on unstratified 3-arms Cox proportional hazard model
Statistical Analysis 6: Comparison: China Nivolumab 240 mg vs China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; China Nivolumab + Ipilimumab over China Nivolumab; Test type: Superiority; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.72 to 2.49] — Hazard Ratios are based on unstratified 3-arms Cox proportional hazard model

5. Secondary Outcome: Overall Survival (OS) in Tumor Mutational Burden (TMB) High and Low Subgroups by TMB Cutoff In The Global Population
Description: Tumor mutational burden (TMB) is measured using FoundationOne CDxTM (F1CDx) assay, a comprehensive genomic profile (CGP) assay based on baseline tumor tissue. TMB is defined as the number of somatic, coding, base substitution, and indel mutations per megabase of genome examined.
  OS in TMB by the following cutoff points: ≥10 mutations/mb, < 10 mutations/mb, ≥13 mutations/mb, <13 mutations/mb
Time Frame: From randomization to the date of death or last known alive date (up to approximately 73 months)
Population: All TMB evaluable participants in the global population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Global Placebo | Global Nivolumab 240 mg | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 192 | 196 | 192
Months
  ≥10 mutations/mb: number analyzed (Participants) | 88 | 98 | 90
  ≥10 mutations/mb | 11.96 [7.49 to 13.67] | 12.81 [9.95 to 18.60] | 10.55 [8.38 to 14.16]
  < 10 mutations/mb: number analyzed (Participants) | 104 | 98 | 102
  < 10 mutations/mb | 9.20 [7.46 to 11.04] | 9.76 [8.34 to 11.30] | 8.11 [6.60 to 10.05]
  ≥13 mutations/mb: number analyzed (Participants) | 59 | 71 | 61
  ≥13 mutations/mb | 9.69 [6.21 to 13.63] | 12.98 [9.95 to 18.60] | 13.47 [9.26 to 21.75]
  <13 mutations/mb: number analyzed (Participants) | 133 | 125 | 131
  <13 mutations/mb | 10.02 [7.66 to 11.47] | 9.89 [8.64 to 11.30] | 7.85 [6.67 to 9.66]
Statistical Analysis 1: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff ≥10 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.61 to 1.15] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 2: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff ≥10 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.55 to 1.04] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 3: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff ≥13 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.42 to 0.92] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 4: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff ≥13 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.44 to 0.93] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 5: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff <10 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.68 to 1.21] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 6: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff <10 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.18] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 7: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff <13 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.81 to 1.35] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 8: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff <13 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.72 to 1.20] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo

6. Secondary Outcome: Progression Free Survival (PFS) Per BICR in Tumor Mutational Burden (TMB) High and Low Subgroups by TMB Cutoff In The Global Population
Description: Tumor mutational burden (TMB) is measured using FoundationOne CDxTM (F1CDx) assay, a comprehensive genomic profile (CGP) assay based on baseline tumor tissue. TMB is defined as the number of somatic, coding, base substitution, and indel mutations per megabase of genome examined.
  PFS in TMB by the following cutoff points: ≥10 mutations/mb, < 10 mutations/mb, ≥13 mutations/mb, <13 mutations/mb.
Time Frame: as for outcome 4
Population: All TMB evaluable participants in the global population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Global Placebo | Global Nivolumab 240 mg | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 192 | 196 | 192
Months
  ≥10 mutations/mb: number analyzed (Participants) | 88 | 98 | 90
  ≥10 mutations/mb | 1.58 [1.41 to 2.63] | 2.79 [2.04 to 4.17] | 2.33 [1.48 to 2.92]
  < 10 mutations/mb: number analyzed (Participants) | 104 | 98 | 102
  < 10 mutations/mb | 1.41 [1.35 to 1.45] | 1.61 [1.45 to 2.53] | 1.48 [1.41 to 2.00]
  ≥13 mutations/mb: number analyzed (Participants) | 59 | 71 | 61
  ≥13 mutations/mb | 1.58 [1.41 to 2.63] | 2.76 [1.61 to 4.11] | 2.63 [1.48 to 3.81]
  <13 mutations/mb: number analyzed (Participants) | 133 | 125 | 131
  <13 mutations/mb | 1.41 [1.38 to 1.45] | 1.84 [1.48 to 2.66] | 1.48 [1.41 to 2.00]
Statistical Analysis 1: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff ≥10 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.58 to 1.09] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 2: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff ≥10 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.50 to 0.92] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 3: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff ≥13 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.50 to 1.07] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 4: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff ≥13 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.46 to 0.95] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 5: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff <10 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.54 to 0.96] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 6: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff <10 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.49 to 0.89] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 7: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; TMB cutoff <13 mutations/mb: Nivo+Ipi over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.60 to 1.01] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo
Statistical Analysis 8: Comparison: Global Placebo vs Global Nivolumab 240 mg; TMB cutoff <13 mutations/mb: Nivo over placebo; Test type: Superiority; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.53 to 0.89] — Unstratified Cox proportional hazard model. Hazard Ratios are experimental treatment group over placebo

7. Post Hoc Outcome: Overall Survival (OS) of Nivolumab + Ipilimumab Versus Placebo - Extended Collection
Description: Overall survival (OS) comparing nivolumab + ipilimumab versus placebo. OS was defined as the time from randomization to the date of death. A participant who had not died was censored at last known alive date. OS was followed up during the blinded study drug treatment and every 3 months via in-person or phone contact after participant discontinued the blinded study drug.
  Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 11-Nov-2021).
Time Frame: From randomization to the date of death or last known alive date (up to approximately 73 months)
Population: All randomized participants in the nivolumab + ipilimumab and placebo arms
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Global Placebo | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | China Placebo | China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
Number analyzed (Participants) | 275 | 279 | 26 | 24
Months | 9.56 [8.18 to 11.01] | 9.17 [8.15 to 10.35] | 9.28 [5.59 to 14.26] | 10.48 [7.13 to 13.40]
Statistical Analysis 1: Comparison: Global Placebo vs Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; Global nivolumab + ipilimumab over Global placebo; Test type: Superiority; Stratified Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.76 to 1.09] — Hazard Ratios are based on stratified 3-arms Cox proportional hazard model
Statistical Analysis 2: Comparison: China Placebo vs China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg; China nivolumab + ipilimumab over China placebo; Test type: Superiority; Stratified Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.52 to 1.67] — Hazard Ratios are based on unstratified 3-arms Cox proportional hazard model

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from randomization until study completion (up to approximately 73 months). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy (up to approximately 34 months).
Description: The total number at risk for all-cause mortality represents all participants who were randomized. The total number at risk by any serious adverse event and other (not including serious) adverse events represents all participants that received at least 1 dose of study medication.
Arm/Group | Global Placebo | Global Nivolumab 240 mg | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg | China Placebo | China Nivolumab 240 mg | China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 250/275 | 231/280 | 240/279 | 24/26 | 23/25 | 23/24
Serious Adverse Events (participants affected / at risk) | 117/273 | 131/279 | 198/278 | 8/26 | 10/25 | 19/24
Other Adverse Events (participants affected / at risk) | 228/273 | 244/279 | 263/278 | 22/26 | 23/25 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Global Placebo (N=273) | Global Nivolumab 240 mg (N=279) | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=278) | China Placebo (N=26) | China Nivolumab 240 mg (N=25) | China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 3 | 7 | 0 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 4 | 0 | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 1 | 3 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Papilloedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 19 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 16 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 5 | 0 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 6 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 2 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 3 | 0 | 1 | 0
Facial pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 7 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 5 | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 3 | 8 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 4 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 3 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 2
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Cytomegalovirus enteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0
Gastric infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infective thrombosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 6 | 12 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 2 | 8 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
General physical condition abnormal (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 2 | 1 | 2 | 0
Transaminases increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 3 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 6 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 7 | 9 | 0 | 1 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 50 | 50 | 51 | 4 | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Metastases to spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Immune-mediated encephalitis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Limbic encephalitis (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Bladder mass (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Immune-mediated cystitis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 3 | 0 | 0 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 4 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 14 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0
Superior vena cava stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 4 | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Global Placebo (N=273) | Global Nivolumab 240 mg (N=279) | Global Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=278) | China Placebo (N=26) | China Nivolumab 240 mg (N=25) | China Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg (N=24)
Anaemia (Blood and lymphatic system disorders) | 31 | 30 | 25 | 10 | 4 | 12
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 4 | 6 | 2 | 3 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 5 | 8 | 6 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4 | 10 | 1 | 0 | 5
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 6 | 18 | 28 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 3 | 23 | 30 | 1 | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 13 | 16 | 22 | 0 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 14 | 10 | 11 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 37 | 34 | 51 | 1 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 47 | 59 | 88 | 2 | 0 | 4
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 67 | 69 | 78 | 3 | 3 | 4
Toothache (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 21 | 27 | 47 | 3 | 0 | 2
Asthenia (General disorders) | 36 | 39 | 45 | 2 | 3 | 0
Chest discomfort (General disorders) | 2 | 2 | 2 | 0 | 0 | 3
Chest pain (General disorders) | 8 | 10 | 9 | 1 | 2 | 1
Fatigue (General disorders) | 66 | 88 | 86 | 2 | 0 | 7
Malaise (General disorders) | 7 | 6 | 9 | 1 | 1 | 7
Non-cardiac chest pain (General disorders) | 17 | 10 | 11 | 3 | 0 | 0
Oedema peripheral (General disorders) | 15 | 16 | 18 | 0 | 1 | 1
Pain (General disorders) | 3 | 7 | 5 | 1 | 2 | 0
Pyrexia (General disorders) | 11 | 20 | 43 | 4 | 3 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 2 | 1 | 0 | 3
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 3 | 2 | 5 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 6 | 15 | 14 | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 13 | 14 | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 8 | 7 | 7 | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 12 | 21 | 43 | 4 | 6 | 11
Amylase increased (Investigations) | 9 | 9 | 19 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 10 | 19 | 39 | 3 | 7 | 10
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 5 | 10 | 12 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 3 | 2 | 3 | 0 | 2 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 9 | 11 | 19 | 1 | 2 | 3
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
Blood urea increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 4 | 8 | 2 | 3 | 2
Lipase increased (Investigations) | 11 | 12 | 28 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 15 | 11 | 10 | 8 | 4 | 4
Platelet count decreased (Investigations) | 5 | 12 | 14 | 3 | 5 | 1
Thyroxine free decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2
Weight decreased (Investigations) | 12 | 16 | 27 | 1 | 0 | 6
White blood cell count decreased (Investigations) | 7 | 8 | 6 | 7 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 57 | 71 | 101 | 8 | 7 | 9
Dehydration (Metabolism and nutrition disorders) | 7 | 10 | 17 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 13 | 19 | 1 | 3 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 5 | 9 | 2 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 5 | 8 | 0 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 11 | 20 | 2 | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 11 | 15 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 22 | 35 | 2 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 35 | 31 | 1 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 30 | 22 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 8 | 13 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 26 | 22 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 24 | 29 | 28 | 0 | 0 | 2
Headache (Nervous system disorders) | 27 | 37 | 49 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 16 | 19 | 25 | 2 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 55 | 53 | 10 | 6 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 64 | 49 | 2 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 4 | 3 | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 13 | 5 | 0 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 11 | 18 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 6 | 7 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 43 | 80 | 0 | 2 | 7
Rash (Skin and subcutaneous tissue disorders) | 16 | 20 | 68 | 0 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 10 | 26 | 0 | 0 | 2
Hypotension (Vascular disorders) | 2 | 7 | 14 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02538666/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT02538666/SAP_001.pdf